CLINICAL TRIAL: NCT00730574
Title: Examining the Commonness of the C677T Mutation in the MTHFR Gene in Subjects With B12 Deficiency and the Influence of the B12 Deficiency Combined With the C677T Mutation on the MTHFR Gene on Endothelial Function.
Brief Title: Examining B12 Deficiency Associated With C677T Mutation on MTHFR Gene in Terms of Commonness and Endothelial Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: completed patient rectuitment
Sponsor: Moshe Flugelman (Other)
Responsible Party: Sponsor-Investigator, Moshe Flugelman, Principal Investigator and Sponsor, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CMC-07-0070-CTIL
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: B12 Deficiency Combined With C677T Mutation on MTHFR Gene
MeSH Terms: interventions — Vitamin B 12; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (No Intervention): The control group, marked B, gets only B12 vitamin 1mg/day treatment to comply with ethics regulations seeing as they do suffer from B12 deficiency .
- A (Experimental): The trial group which receives daily treatment of 1mg Vitamin B12 (sublingual tablets) combined with 5 mg Folic acid (tablets)
  Interventions: Dietary Supplement: Vitamin B12 + Folic Acid

INTERVENTIONS:
Dietary Supplement: Vitamin B12 + Folic Acid — Trial group would get daily treatment of 1 mg Vitamin B12 combined with 5 mg Folic Acid
  Other Names: Vitamin B12, 1 mg, by Solgar; Folic acid, 5 mg, by Rakah
  Arms: A

SUMMARY:
The purpose of this study is to determine the commonness of the C677T mutation in the MTHFR gene in subjects with B12 deficiency. Also, we'd like to investigate the effect of B12 deficiency combined with the C677T mutation on endothelial function.

DETAILED DESCRIPTION:
we showed that patiebts with B12 deficiency have higher than expected frequency of MTHFR mutation and patients with both abnormalities havean abnormal endothelial function

ELIGIBILITY:
Inclusion Criteria:

1. adult males and females of the broad population aged 20-60
2. with no symptomatic heart disease/condition
3. with Vitamin B12 levels of 150 pmol or less
4. which have not received Vitamin B12 supplement treatment before

Exclusion Criteria:

1. Adults suffering from a known heart disease/condition
2. any disease the investigator might find as interfering with the process of the experiment
3. tumor-oriented diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary measure to determine the effect of the treatment will be reduced levels of Homocysteine in subjects with B12 deficiency combined with C677T mutation in the MTHFR gene. | The key measure would be measured upon enrollment and 6 weeks afterwards, upon completion of treatment based on 1mg Vitamin B12 sublinual and 5 mg Folic Acid per day.

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Y Flugelman, Principal Investigator — Carmel Medical Center, Haifa, Israel
Locations (1):
- Carmel Medical Center, Haifa, Israel